CLINICAL TRIAL: NCT02727907
Title: International, Multicenter, Double-blinded, Placebo-controlled, Randomized Study of the Efficacy and Safety of Drugs BCD-033 and Rebif for the Treatment of Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Study of Efficacy and Safety of Drugs BCD-033 and Rebif for Treatment of Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BCD-033-2
Record Dates: First submitted 2015-05-29; First posted 2016-04-05 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCD-033 (Experimental): Subcutaneous injection of BCD-033, 44 µg (0,5 ml) 3 times per week, every other day, for 92 weeks
  Interventions: Drug: BCD-033 (interferon beta 1a)
- Rebif (Active Comparator): Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks, followed by 48 weeks of open-label BCD-033 usage
  Interventions: Drug: Rebif (interferon beta 1a)
- Placebo (Placebo Comparator): Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for 48 weeks, followed by 72 weeks of open-label BCD-033 usage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCD-033 (interferon beta 1a) — Subcutaneous injection of BCD-033, 44 µg (0,5 ml) 3 times per week, every other day, for 92 weeks
  Arms: BCD-033
Drug: Rebif (interferon beta 1a) — Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks
  Arms: Rebif
Drug: Placebo — Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for12 weeks
  Arms: Placebo

SUMMARY:
Study design is double-blind, randomized, placebo-controlled study in 3 parallel groups with the use of active comparator and placebo. Total duration of therapy of about 2 years. Study hypothesis is equivalence of efficacy and safety of the investigational drug BCD-033 original drug Rebif®.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. Patients of both genders with Multiple Sclerosis (McDonald criteria 2010)
3. No relapses 28 days before randomisation
4. Expanded Disability Status Scale score 0-5,5

Exclusion Criteria

1. Primary or secondary progression of Multiple Sclerosis
2. Expanded Disability Status Scale score more then 5,5
3. Severe depression, suicide ideas and/or attempts
4. Systemic corticosteroid application in 30 days before randomisation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific neurology center, RAS, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-033: Subcutaneous injection of BCD-033, 44 µg (0,5 ml) 3 times per week, every other day, for 96 weeks BCD-033 (interferon beta 1a): Subcutaneous injection of BCD-033, 44 µg (0,5 ml) 3 times per week, every other day, for 96 weeks
- Rebif/BCD-033: Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks, followed by 48 weeks of open-label BCD-033 usage Rebif (interferon beta 1a): Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks
- Placebo/BCD-033: Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for 16 weeks, followed by 68 weeks of open-label BCD-033 usage
Period: Overall Study
Arm/Group | BCD-033 | Rebif/BCD-033 | Placebo/BCD-033
Started | 53 | 56 | 54
Recived One Injection of Drug | 53 | 55 | 54
Completed | 40 | 43 | 43
Not Completed | 13 | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- BCD-033: interferon beta-1a (BCD-033)
- Rebif / BCD-033: interferon beta-1a (Rebif / BCD-033)
- Placebo / BCD-033: placebo / interferon beta-1a
- Total: Total of all reporting groups
Arm/Group | BCD-033 | Rebif / BCD-033 | Placebo / BCD-033 | Total
Number analyzed (Participants) | 53 | 55 | 54 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 55 | 54 | 162
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28.00 [25.00 to 39.0] | 30.00 [26.0 to 37.0] | 29.5 [26.0 to 38.0] | 29.0 [26.0 to 38.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 31 | 34 | 103
  Male | 15 | 24 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Combined Unique Active Lesions
Description: Number of Combined Unique Active Lesions (CUA) -- the number of new MRI contrast uptake lesions on T1 images, and new or expanding lesions on T2 images (lesion identified on T1-and T2 images is not counted twice) after 52 weeks blinded application of interferon-β1а (BCD-033 and Rebif®) (44 mcg).
Time Frame: 52 weeks
Population: The primary endpoint was assessed after 52 weeks of use of IFN-β1a (BCD-033 and Rebif) in a full dose (44 μg). In the analysis of the effeciency of MRI indicators included 100 patients
Measure: Median (Inter-Quartile Range); unit: lesions
Groups:
- Rebif: Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks, followed by 48 weeks of open-label BCD-033 usage Rebif (interferon beta 1a): Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks
Arm/Group | BCD-033 | Rebif
Number analyzed (Participants) | 44 | 46
lesions | 0.0 [0.0 to 1.25] | 0.0 [0.0 to 1.0]

2. Secondary Outcome: Annual Relapse Rate
Description: Annual relapse rate ARR for 52 weeks was evaluated in all three groups, after the application of IFN beta-1a
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: relapses
Groups:
- Rebif / BCD-033: Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks, followed by 48 weeks of open-label BCD-033 usage Rebif (interferon beta 1a): Subcutaneous injection of Rebif, 44 µg (0,5 ml) 3 times per week, every other day, for 48 weeks
- Placebo / BCD-033: Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for 16 weeks, followed by 68 weeks of open-label BCD-033 usage
Arm/Group | BCD-033 | Rebif / BCD-033 | Placebo / BCD-033
Number analyzed (Participants) | 53 | 55 | 55
relapses | 0.113 (0.375) | 0.091 (0.348) | 0.109 (0.369)

3. Secondary Outcome: Proportion of Subjects Without Confirmed Relapse
Description: proportion of subjects without confirmed relapse in PP
Time Frame: 16, 52 weeks
Population: The analysis was performed in per protocol population at 16 and 52 weeks
Measure: Number; unit: Count of Participants
Groups:
- Placebo: Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for 16 weeks, followed by 68 weeks of open-label BCD-033 usage
Arm/Group | BCD-033 | Rebif | Placebo
Number analyzed (Participants) | 53 | 51 | 51
Count of Participants
  week 16 | 49 | 46 | 45
  week 52: number analyzed (Participants) | 46 | 48 | 43
  week 52 | 41 | 44 | 39

4. Secondary Outcome: Relapse Free Time
Description: Time to first relapse in "per protocol" population
Time Frame: 96 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 40 | 45
days | 207.0 [52.0 to 276.0] | 183.0 [26.0 to 286.0]

5. Secondary Outcome: Number of Combined Unique Active Lesions
Description: CUA (the number of new contrast-enhanced lesions on T1 images, and new or expanding lesions on T2 images (lesion identified on T1-and T2 images is not counted twice)
Time Frame: 96 weeks
Measure: Median (Inter-Quartile Range); unit: lesions
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 44 | 46
lesions | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

6. Secondary Outcome: Annual Relapse Rate
Description: Annual Relapse Rate ARR for 96 weeks was evaluated in two groups, after the administraion of IFN beta-1a in a full dose for 96 weeks.
Time Frame: 96 week
Measure: Mean (Standard Error); unit: relapses
Arm/Group | BCD-033 | Rebif
Number analyzed (Participants) | 53 | 55
relapses | 0.208 (0.532) | 0.145 (0.524)

7. Secondary Outcome: Relapse Free Time
Description: Time to first relapse in "per protocol" population
Time Frame: 16, 52 weeks
Population: The analysis was performed in per protocol population at 16 and 52 weeks
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Placebo/BCD-033: Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for 48 weeks, followed by 72 weeks of open-label BCD-033 usage
  Placebo: Subcutaneous injection of placebo, 0,5 ml 3 times per week, every other day, for12 weeks
Arm/Group | BCD-033 | Rebif | Placebo/BCD-033
Number analyzed (Participants) | 53 | 51 | 51
days
  week 16 | 33.5 [12.0 to 60.0] | 14.0 [12 to 26.0] | 15.0 [5.0 to 61.75]
  week 52: number analyzed (Participants) | 46 | 48 | 51
  week 52 | 193.0 [51.5 to 240.0] | 123.5 [22.5 to 204.75] | 74.0 [25.0 to 210.0]

8. Secondary Outcome: Number of Combined Unique Active Lesions
Description: as for outcome 5
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: lesions
Arm/Group | BCD-033 | Rebif | Placebo
Number analyzed (Participants) | 53 | 51 | 51
lesions | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0] | 1.0 [0.0 to 3.0]

9. Other Pre Specified Outcome: Adverse Events/Serious Adverse Events
Description: quantity and grade of all AE/SAE is calculated in subjects, who received at least one dose of study drug
Time Frame: 96 weeks
Measure: Number; unit: adverse events
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 53 | 55
adverse events | 124 | 110

10. Other Pre Specified Outcome: Severe Adverse Events Frequency
Description: AE grade 3-4 (CTCAE 4.03) is calculated in subjects, who received at least one dose of study drug
Time Frame: 52 weeks
Measure: Number; unit: adverse events
Arm/Group | BCD-033 | Rebif | Placebo/BCD-033
Number analyzed (Participants) | 53 | 55 | 54
adverse events | 5 | 4 | 7

11. Other Pre Specified Outcome: Withdrawal
Description: quantity of withdrawals due to AE/SAE is calculated in subjects, who received at least one dose of study drug
Time Frame: 16, 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-033 | Rebif | Placebo/BCD-033
Number analyzed (Participants) | 53 | 55 | 54
Participants
  week 16 | 0 | 1 | 1
  week 52 | 1 | 1 | 2

12. Other Pre Specified Outcome: Immunogenicity
Description: Count of Participants with Binding and Neutralizing Antibodies
Time Frame: 16, 52 weeks
Measure: Number; unit: participants
Arm/Group | BCD-033 | Rebif/BCD-033 | Placebo/BCD-033
Number analyzed (Participants) | 51 | 49 | 53
participants
  week 16 : Binding Antibodies | 6 | 5 | 2
  week 16 : Neutralizing Antibodies | 5 | 5 | 2
  week 52 : Binding Antibodies | 10 | 9 | 7
  week 52 : Neutralizing Antibodies | 9 | 8 | 7

13. Other Pre Specified Outcome: Adverse Reaction/Serious Adverse Reactions
Description: quantity and grade of all adverse reactions/serious adverse reactions is calculated in subjects, who received at least one dose of study drug
Time Frame: 16, 52 weeks
Measure: Number; unit: adverse events
Arm/Group | BCD-033 | Rebif | Placebo/BCD-033
Number analyzed (Participants) | 53 | 55 | 54
adverse events
  week 16 | 67 | 59 | 33
  week 52 | 92 | 80 | 92

14. Other Pre Specified Outcome: Severe Adverse Events Frequency
Description: AE grade 3-4 (CTCAE 4.03)is calculated in subjects, who received at least one dose of study drug
Time Frame: 96 weeks
Measure: Number; unit: adverse events
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 53 | 55
adverse events | 2 | 3

15. Other Pre Specified Outcome: Withdrawal
Description: quantity of withdrawals due to AE/SAE is calculated in subjects, who received at least one dose of study drug
Time Frame: 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 53 | 55
Participants | 1 | 1

16. Other Pre Specified Outcome: Immunogenicity
Description: Count of Participants with Binding and Neutralizing Antibodies
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | BCD-033 | Rebif/BCD-033
Number analyzed (Participants) | 51 | 49
participants
  Binding Antibodies | 19 | 14
  Neutralizing Antibodies | 16 | 13

17. Other Pre Specified Outcome: Serious Adverse Events
Description: quantity and grade of all SAE is calculated in subjects, who received at least one dose of study drug
Time Frame: 52 week of study
Measure: Number; unit: adverse events
Arm/Group | BCD-033 | Rebif/BCD-033 | Placebo/BCD-033
Number analyzed (Participants) | 53 | 55 | 54
adverse events | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: 52 week
Arm/Group | BCD-033 | Rebif | Placebo/BCD-033
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/55 | 2/54
Other Adverse Events (participants affected / at risk) | 35/53 | 32/55 | 34/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-033 (N=53) | Rebif (N=55) | Placebo/BCD-033 (N=54)
nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — The patient had an albuminuria, in connection with which he was hospitalized in a hospital for treatment. It is discharged with improvement of a status. The therapy was abolished.
Left hemophthalmos (Eye disorders) | NA | NA | 1 (1)
Chronic viral hepatitis B (Infections and infestations) | NA | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-033 (N=53) | Rebif (N=55) | Placebo/BCD-033 (N=54)
headache (General disorders) | 3 | 3 | 3
flu-like syndrom (General disorders) | 15 | 16 | 19
fever (General disorders) | 7 | 6 | 6
increased ALT (Investigations) | 3 | 4 | 3
local reaction (General disorders) | 15 | 12 | 10
lymphopenia (Investigations) | 5 | 4 | 4
neutropenia (Investigations) | 11 | 4 | 10
thrombocytopenia (Investigations) | 3 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No